CLINICAL TRIAL: NCT03804359
Title: Personalized Medicine for Membranous Nephropathy
Acronym: PMMN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-APN-01
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: Nephrotic Syndrome; PLA2R1-antibodies; Epitope spreading; Rituximab
MeSH Terms: conditions — Glomerulonephritis, Membranous; Nephrotic Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEMRITUX protocol (No Intervention): 6 months of symptomatic antihypertensive and antiproteinuric therapy, and if the nephrotic syndrome persists at month-6 (urinary protein/creatinine ratio (UPCR) remains > 3.5 g/g and albuminemia < 30 g/l), two 375 mg/m2 rituximab infusions at 1-week interval.
- Personalized treatment (Experimental): * restricted anti-CysR activity at inclusion : 6-month symptomatic antihypertensive and antiproteinuric treatment (KDIGO)
  * restricted anti-CysR activity after 6 months of symptomatic treatment with persisting nephrotic syndrome (UPCR remains > 3.5 g/g and albuminemia < 30 g/l): two 375 mg/m2 rituximab infusions at 1-week interval;
  * Anti-CTLD1/7 activity at inclusion or after 6 months with persisting nephrotic syndrome (UPCR remains > 3.5 g/g and albuminemia < 30 g/l): two 1g rituximab infusions at 2-week interval at month 0 and/or month 6.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — In the "personalized arm", the patient will be treated in function of the CysR activity result during the inclusion visit.
  Arms: Personalized treatment

SUMMARY:
Randomized, open label, multicentre (20 sites), prospective trial comparing the efficacy of two therapeutic strategies to obtain clinical remission 1 year after diagnosis of Idiopathic Membranous Nephropathy with nephrotic syndrome and anti-PLA2R1 (phospholipase A2 receptor 1) antibodies:

* GEMRITUX protocol: 6 months of symptomatic antihypertensive and antiproteinuric therapy, and if the nephrotic syndrome persists at month-6 (urinary protein/creatinine ratio (UPCR) remains > 3.5 g/g and albuminemia < 30 g/l), two 375 mg/m2 rituximab infusions at 1-week interval.
* Personalized treatment:

  * restricted anti-CysR activity at inclusion : 6-month symptomatic antihypertensive and antiproteinuric treatment (KDIGO)
  * restricted anti-CysR activity after 6 months of symptomatic treatment with persisting nephrotic syndrome (UPCR remains > 3.5 g/g and albuminemia < 30 g/l): two 375 mg/m2 rituximab infusions at 1-week interval;
  * Anti-CTLD (C-type lectin domains ) 1/7 activity at inclusion or after 6 months with persisting nephrotic syndrome (UPCR remains > 3.5 g/g and albuminemia < 30 g/l): two 1g rituximab infusions at 2-week interval at month 0 and/or month 6.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Anti-PLA2R1 activity detected by ELISA or Euroimmune Immunofluorescence Assay
* Nephrotic syndrome defined by proteinuria > 3.5 g/24h (or UPCR > 3.5 g/g) and serum albumin < 30 g/L at diagnosis
* eGFR (CKD-EPI) > 30 ml/min/1,73 m2 at diagnosis
* Symptomatic treatment according to KDIGO guidelines: maximal tolerated dose of NIAT : Non Immunosuppressive Antiproteinuric Treatment (angiotensin-converting enzyme inhibitor and/or angiotensin 2 receptor blockers, diuretics and statins)
* Medical insurance
* Signed informed consent
* Having understood and accepted the need for long-term medical follow-up
* Woman of child-bearing age must be using an effective method of contraception

Exclusion Criteria:

* Secondary Membranous Nephropathy: Membranous Nephropathy related to cancer, infectious, systemic lupus erythematosis, drug
* Anti-PLA2R1 antibodies not confirmed by central analysis (in this case the patient will be replaced)
* Pregnancy or breastfeeding
* Immunosuppressive treatment in the 3 last months
* Cancer under treatment
* Patient with complicated nephrotic syndrome that would require early immunosuppressive treatment (thrombosis, acute renal failure…)
* Patients with active, severe infections or active hepatitis B
* Hypersensitivity to the active substance or to murine proteins, or to any of the other excipients
* Patients in a severely immunocompromised state
* Severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease
* Patients unable to give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Clinical remission will be defined as a composite criterion combining (KDIGO definitions) | 6 months
  * Complete clinical remission: urinary protein/creatinine ratio (UPCR)<0.3 g/g in spot morning urine samples and serum albumin > 35 g/L and eGFR (epidermal growth factor receptor) > 60 ml/min/1.73 m2
  * Partial clinical remission: UPCR < 3.5 g/g with a decrease greater than 50% from baseline and serum albumin > 30 g/L and increase of serum creatinine lower than 20%

SECONDARY OUTCOMES:
Immunological remission | 6 months
  full PLA2R1 depletion measured by ELISA (titer<14RU (relative units) /ml)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara SEITZ-POLSKI, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (19):
- France (19):
  - CHU D'amiens Hôpital Sud, Amiens
  - CHU Besançon, Besançon
  - Hôpital universitaire La Cavale Blanche, Brest
  - CHU de Caen, Caen
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - CHRU de LILLE, Lille
  - CHU de LYON NORD, Lyon
  - AP-HM, Marseille
  - CHRU de Montpellier, Montpellier
  - CHU de NANTES, Nantes
  - Dr Barbara SEITZ-POLSKI, Nice
  - CHU Carémeau, Nîmes
  - Hôpital Necker, Paris
  - Le Kremlin Bicêtre, Paris
  - Hôpital de la maison blanche, Reims
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours

REFERENCES:
- [Background] Simon N, Courouce AM, Lemarrec N, Trepo C, Ducamp S. A twelve year natural history of hepatitis C virus infection in hemodialyzed patients. Kidney Int. 1994 Aug;46(2):504-11. doi: 10.1038/ki.1994.301. PMID 7967364
- [Background] Simon P, Ramee MP, Boulahrouz R, Stanescu C, Charasse C, Ang KS, Leonetti F, Cam G, Laruelle E, Autuly V, Rioux N. Epidemiologic data of primary glomerular diseases in western France. Kidney Int. 2004 Sep;66(3):905-8. doi: 10.1111/j.1523-1755.2004.00834.x. PMID 15327379
- [Background] Ponticelli C. Membranous nephropathy. J Nephrol. 2007 May-Jun;20(3):268-87. PMID 17557260
- [Background] Glassock RJ. The pathogenesis of idiopathic membranous nephropathy: a 50-year odyssey. Am J Kidney Dis. 2010 Jul;56(1):157-67. doi: 10.1053/j.ajkd.2010.01.008. Epub 2010 Apr 8. PMID 20378220
- [Result] Lassalle M, Ayav C, Frimat L, Jacquelinet C, Couchoud C; Au Nom du Registre REIN. The essential of 2012 results from the French Renal Epidemiology and Information Network (REIN) ESRD registry. Nephrol Ther. 2015 Apr;11(2):78-87. doi: 10.1016/j.nephro.2014.08.002. Epub 2014 Nov 1. PMID 25457107
- [Derived] Brglez V, Boyer-Suavet S, Zorzi K, Fernandez C, Fontas E, Esnault V, Seitz-Polski B. Personalized Medicine for PLA2R1-Related Membranous Nephropathy: A Multicenter Randomized Control Trial. Front Med (Lausanne). 2020 Aug 13;7:412. doi: 10.3389/fmed.2020.00412. eCollection 2020. PMID 32903623